CLINICAL TRIAL: NCT03210948
Title: Conventional Versus Elastography Targeted Endoscopic Ultrasound Fine Needle Aspiration of Solid Pancreatic Lesions: a Randomized Controlled Trial
Brief Title: Conventional Versus Elastography Targeted Endoscopic Ultrasound Fine Needle Aspiration of Solid Pancreatic Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ospedali Riuniti di Foggia (Other)
Responsible Party: Principal Investigator, Antonio Facciorusso, MD, Ospedali Riuniti di Foggia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: EUS01
Record Dates: First submitted 2017-07-04; First posted 2017-07-07 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RTE-guided EUS-FNA (Experimental): The needle will be then inserted into the most suspicious part ("dark blue") of the lesion as assessed at real time elastography.
  Interventions: Device: RTE-guided EUS-FNA
- Conventional EUS-FNA (Active Comparator): A 25 G needle with a central stylet to protect the aspiration channel of the needle will be introduced though the endoscope's working channel.
  Interventions: Device: Conventional EUS-FNA

INTERVENTIONS:
Device: RTE-guided EUS-FNA — Fine needle aspiration with 25 gauge needle under RTE-guidance
  Arms: RTE-guided EUS-FNA
Device: Conventional EUS-FNA — Fine needle aspiration with no RTE guidance
  Arms: Conventional EUS-FNA

SUMMARY:
Diagnostic assessment of solid pancreatic lesions may represent a real challenge in the clinical practice, even with the aid of tissue sampling by means of endoscopic ultrasound (EUS) fine needle aspiration (FNA).

Aim of this randomized controlled trial (RCT) is to establish the diagnostic accuracy, sensitivity, and specificity of real time elastography (RTE)-guided EUS-FNA as compared to conventional EUS-FNA in a series of patients with solid pancreatic masses.

Eligible will be patients with solid pancreatic masses detected at abdominal imaging (ultrasound, CT-scan or MRI).

In the treatment arm, RTE assessment of pancreatic masses will be performed using a last generation ultrasound machine, and all suspicious areas at elastography (i.e. those appearing in dark blue color as a consequence of higher cellularity of tumoral tissue) will be recorded and stored in our database. A 25 G needle will be then inserted into the most suspicious part ("dark blue") of the lesion and immediately after the procedure the stylet will be removed. At the end of the procedure, the needle will be retracted and the samples will be prepared for cytological examination.

Primary endpoint will be diagnostic yield of the procedure. Secondary endpoints the diagnostic sensitivity, specificity, number of passes needed to achieve an adequate sample and safety It will be planned to enroll 142 patients (71 per arms) within 1 year. A minimum follow up of 6 months from the last patient unsuitable to surgery will be required.

DETAILED DESCRIPTION:
To establish the diagnostic accuracy, sensitivity, and specificity of RTE-guided EUS-FNA as compared to conventional EUS-FNA in a series of patients with solid pancreatic masses.

Protocol design Phase II, two-arms, open-label, randomized controlled trial.

Trial population Patients with solid pancreatic masses detected at abdominal imaging (ultrasound, CT-scan or MRI).

Protocol Treatments

* The Treatment arm will undergo RTE-guided EUS-FNA with 25 G needle.
* The Control arm will undergo conventional EUS-FNA with 25 G needle.

Technical procedure

Under sedation with propofol, EUS will be performed using a curved-array transducer. A 25 G needle with a central stylet to protect the aspiration channel of the needle will be introduced though the endoscope's working channel. RTE assessment of pancreatic masses will be performed using a last generation ultrasound machine, and all suspicious areas at elastography (i.e. those appearing in dark blue color as a consequence of higher cellularity of tumoral tissue) will be recorded and stored in our database. Beside qualitative assessment based on red-green-blue color map, a semi-quantitative approach providing a numeric value expressed as strain ratio5 will be undertaken.

The needle will be then inserted into the most suspicious part ("dark blue") of the lesion and immediately after the procedure the stylet will be removed. More than 10 to- and fro- movements will be made within the lesion and aspiration will be obtained with a 10 cm3 suction syringe applied to the hub of FNA device. Up to four passes will be performed. At the end of the procedure, the needle will be retracted and the samples fixed in 95% ethanol solution. After being grossly checked for adequacy samples will be prepared for cytological examination with Papanicolaou staining.

The reference standard for classification will be surgery or death from PC in those subjects unsuitable to surgery. In particular, if after a follow-up of 6 months there will be no sign of disease progression or if disease regression will be registered, the lesion will be classified as inflammatory.

Lesions diagnosed as malignant by cytopathology on EUS-FNA sample and finally confirmed by surgery or clinical course will be considered to be true positives (TPs); similarly, benign aspirates finally diagnosed as benign will be considered to be true negatives (TNs). On the other hand, those aspirates apparently benign at cytopathological examination which will be finally diagnosed as malignant will be considered to be false negatives (FNs). Non-diagnostic/inconclusive samples will be registered as such in the database and for analytical purposes when computing diagnostic accuracy will be classified as FNs.

Primary Endpoint Diagnostic yield of the procedure.

Secondary Endpoints

* Diagnostic sensitivity
* Diagnostic specificity
* Number of passes needed to achieve an adequate sample
* Safety

Sample size and study duration It will be planned to enroll 142 patients (71 per arms) within 1 year. A minimum follow up of 6 months from the last patient unsuitable to surgery will be required.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid pancreatic masses detected at abdominal imaging (ultrasound, CT-scan or MRI).

Exclusion Criteria:

* Age under 18 years
* Cystic pancreatic lesions
* Lesions < 1 cm
* History of previous gastrectomy
* Patients with severe coagulopathy or under anticoagulant/antiaggregant therapy which could not be suspended
* Refusal to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2019-01-23 (Estimated); Primary Completion 2019-02-20 (Estimated); Study Completion 2019-02-20 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 12 months
  Proportion of correctly classified subjects (true positives+true negatives) among all subjects (true positives+true negatives+false positives+false negatives)

SECONDARY OUTCOMES:
Diagnostic sensitivity | 12 months
  Proportion of subjects with the disease with positive test result in a total group of subjects with the disease
Diagnostic specificity | 12 months
  Proportion of subjects without the disease with negative test result in total of subjects without disease
Number of passes needed to achieve an adequate sample | 1 day
  Number of needle injections into the lesion needed to obtain an adequate and diagnostic sample
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 week
  Side effects

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Facciorusso, MD, Study Director — Ospedali Riuniti di Foggia
Locations (1):
- Ospedali Riuniti Foggia, Foggia, Italy

IPD SHARING:
Plan to Share IPD: No